CLINICAL TRIAL: NCT01223248
Title: A Phase III Randomized Study Comparing Two Dosing Schedules for Hypofractionated Image-Guided Radiation Therapy in Patients With Metastatic Cancer
Brief Title: Randomized Study Comparing Two Dosing Schedules for Hypofractionated Image-Guided Radiation Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Pisa (Other); University of California, San Francisco (Other); The Champalimaud Centre, Lisbon, Portugal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-154
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Melanoma; Ovarian Cancer; Sarcoma; Bone; CNS-Spinal CD/MEMBR, NOS; Lymph Nodes; Soft Tissue
Keywords: radiation; Hypofractionated Image- Guided; IGIMRT; RT; 10-154
MeSH Terms: conditions — Melanoma; Ovarian Neoplasms; Sarcoma; Pyloric Stenosis, Hypertrophic

ARMS (2):
- stereotactic IGIMRT using a single dose of 24 Gy (Experimental): This is a phase III, multicenter, randomized, study comparing two dosing schedules for hypofractionated image-guided radiation therapy to bone, spine, soft tissue, and lymph nodes in patients with metastatic disease
  Interventions: Radiation: IGIMRT using a single dose of 24 Gy
- stereotactic IGIMRT 27 Gy in 3 fractions (Experimental): This is a phase III, multicenter, randomized, study comparing two dosing schedules for hypofractionated image-guided radiation therapy to bone, spine, soft tissue, and lymph nodes in patients with metastatic disease
  Interventions: Radiation: IGIMRT 27 Gy in 3 fractions

INTERVENTIONS:
Radiation: IGIMRT using a single dose of 24 Gy — Pts in both the hypofractionated & single dose arms will receive the same following standard procedures. The only difference between the arms is the dose delivered at each treatment. 20 MSKCC pts (10 per treatment arm) will be accrued to undergo baseline DW-MRI & DCE-MRI pretreatment for both arms & 1 hour after their initial treatment for single fraction pts, & within one hour of their initial & final radiation treatment for the hypofractionated pts. Pts will be considered for this scan based on compliance to scan schedule & MRI availability for performing the scan within one hour of the planned IGRT. 24 MSKCC pts (12 per treatment arm) will be accrued for the blood collection (optional) up to 4 hours prior, 50-90 minutes after, & approximately 24 hours [MCPG2.3]after treatment for single fraction pts. For pts partaking in both sub-studies, the post-treatment blood collection may be done in a 50-120 minute window to account for scheduling conflicts with the research MRI.
  Arms: stereotactic IGIMRT using a single dose of 24 Gy
Radiation: IGIMRT 27 Gy in 3 fractions — Pts in both the hypofractionated & single dose arms will receive the same following standard procedures. The only difference between the arms is the dose delivered at each treatment. 20 MSKCC pts (10 per treatment arm) will be accrued to undergo baseline DW-MRI & DCE-MRI pretreatment for both arms & within 1 hour after their initial treatment for single fraction pts, & within one hour of their initial & final radiation treatment for the hypofractionated pts. Pts will be considered for this scan based on compliance to scan schedule & MRI availability for performing the scan within one hour of the planned IGRT. 24 MSKCC pts (12 per treatment arm) will be accrued for the blood collection (optional) up to 4 hours prior, 50-90 minutes after, & approximately 24 hours [MCPG2.3]after treatment for single fraction pts. For pts partaking in both sub-studies, the post-treatment blood collection may be done in a 50-120 minute window to account for scheduling conflicts with the research MRI.
  Arms: stereotactic IGIMRT 27 Gy in 3 fractions

SUMMARY:
The purpose of this study is to find out which way of giving high-dose radiation works best for treatment of cancer that has spread to bone, the spine, soft tissue, or lymph nodes. This study will look at the effects, good and/or bad, of giving 27 Gy in three fractions (3 days) or 24 Gy in one fraction (1 day) using image-guided intensity-modulated radiotherapy (IG-IMRT). IG-IMRT is radiation that is given directly to the cancer site and reduces the exposure to normal tissue. Currently there are no studies that compare the effects of giving radiation in either hypofractionated doses (higher total doses of radiation spread out over several treatment days) or a single-fraction dose (entire radiation dose given in one treatment session).

The patient may be asked to participate in an additional part of this study where we will get a a (DW/DCE) MRI before treatment start and within one hour after radiation treatment. If the patient is asked to take part in this portion of the study, all they will need to do is get up to 3 MRIs with standard contrast injection. The purpose of this is to see if as a result of the treatment there are changes in the blood flow going to the cancer which could suggest that the treatment may be successful.

In addition some patients can present new lesions and may be asked if they would like to have these new lesions treated on the protocol. If they are given this option, this will not extend their follow up period. The follow up of the new lesions will match with the prior follow up dates.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of cancer (including epithelial carcinoma, sarcoma, and melanoma) The diagnosis can be done at MSKCC or at participating institutions.
* Sites of metastatic disease to be treated on protocol are limited to bone, spine, soft tissue, and lymph nodes only.
* Patients with American Joint Committee on Cancer (6th edition, 2002) Stage IV cancer with distant metastases
* Age 18 years or older
* Life expectancy >3 months
* Maximum tumor dimension of ≤6 cm in lymph nodes, soft tissue, osseous metastases, or spinal metastases seen on imaging (computed tomography [CT], magnetic resonance imaging [MRI], or PET/CT) and considered amenable for RT.
* If the lesion(s) to be treated are soft-tissue or lymph Nodes unidimensionally measurable disease is required. Bone & spine lesions are eligible even if considered non-measurable.
* Measurable disease is defined as:
* ≥ 10mm for soft-tissue lesions
* ≥ 15mm on the short axis of lymph nodes
* KPS ≥ 80
* Patients must have normal bone marrow function as defined below:(within 2 months of registration) Hemoglobin ≥9.0 g/dl Absolute neutrophil count (ANC) ≥1,500/μl Platelets ≥100,000/μl

Exclusion Criteria:

* Prior radiotherapy delivered to the target region
* Disease to be treated on protocol is less than 2 mm from the spinal cord and therefore will not meet dose constraints*
* Pregnancy or Breast-Feeding (Participants of child-bearing potential are eligible but must consent to using effective contraception during therapy and for at least 3 months after completing therapy).
* Chemotherapy given on the day of the planned radiotherapy treatment
* Lesions which comprise >70% of the width of weight bearing bones, such as the femur.
* Existing cortical bone destruction, where orthopedic stabilization would be required.
* Areas to be treated on protocol do not include metastases to liver, brain or lung.

  * Note: Patients with eligible and ineligible lesions will be accrued to this protocol. Only target eligible lesions will be treated per protocol. Other eligible and ineligible lesions will be treated at the discretion of the treating physician."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To compare the loco-regional control rates of two established hypo-fractionated radiation treatment regimens | 2 years
  a single dose of 24 Gy versus 27 Gy in three fractions for patients with metastatic disease

SECONDARY OUTCOMES:
To compare toxicity outcomes | 2 years
To compare patterns of failure between these two cohorts. | 2 years
To look at changes in SUV uptake as a measure of tumor response. | 2 years
  For patients who are followed with PET/CTs
changes in tumor perfusion | 2 years
  resulting from high-dose IGRT for patients treated with this approach to focal metastases using dynamic contrast-enhanced (DCE)-MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiya Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
- University of Pisa, Pisa, Italy
- The Champalimaud Centre, Lisbon, Portugal

REFERENCES:
- [Derived] Zelefsky MJ, Yamada Y, Greco C, Lis E, Schoder H, Lobaugh S, Zhang Z, Braunstein S, Bilsky MH, Powell SN, Kolesnick R, Fuks Z. Phase 3 Multi-Center, Prospective, Randomized Trial Comparing Single-Dose 24 Gy Radiation Therapy to a 3-Fraction SBRT Regimen in the Treatment of Oligometastatic Cancer. Int J Radiat Oncol Biol Phys. 2021 Jul 1;110(3):672-679. doi: 10.1016/j.ijrobp.2021.01.004. Epub 2021 Jan 8. PMID 33422612
- [Derived] Bodo S, Campagne C, Thin TH, Higginson DS, Vargas HA, Hua G, Fuller JD, Ackerstaff E, Russell J, Zhang Z, Klingler S, Cho H, Kaag MG, Mazaheri Y, Rimner A, Manova-Todorova K, Epel B, Zatcky J, Cleary CR, Rao SS, Yamada Y, Zelefsky MJ, Halpern HJ, Koutcher JA, Cordon-Cardo C, Greco C, Haimovitz-Friedman A, Sala E, Powell SN, Kolesnick R, Fuks Z. Single-dose radiotherapy disables tumor cell homologous recombination via ischemia/reperfusion injury. J Clin Invest. 2019 Feb 1;129(2):786-801. doi: 10.1172/JCI97631. Epub 2019 Jan 14. PMID 30480549
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm